CLINICAL TRIAL: NCT03728270
Title: Assessment of Maximal Incisal Opening Using Patient Specific Titanium Eminoplasty Versus Inlay Autogenous Bone Graft for Treatment of Chronic Mandibular Condylar Dislocation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rania Ihab Younis, Assistant Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 33377576
Record Dates: First submitted 2018-10-25; First posted 2018-11-02 (Actual); Last update posted 2018-11-02 (Actual); Status verified 2018-10

CONDITIONS: Chronic Mandibular Condylar Dislocation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Patient Specific Titanium Eminoplasty (Experimental): * The stages of virtual surgical planning and fabrication of patient specific titanium eminoplasty will be designed my Mimics 15 program.
  * Once designed, the virtual design and surgery will be planned on a computer model where vital anatomical structures could be identified and thus could be avoided during surgery.
  * After obtaining all the dataset needed from the CT scan, the collected data will be sent to the Egyptian soil, water and environmental institution for manufacturing, packing and sterilization of the patient specific titanium eminence.
  * The patient specific titanium eminence will be inserted and secured with two to three screws of individual lengths according to the virtual plan.
  * Functional mandibular movements were reproduced to confirm absence of subluxation and checked for interference and any required adjustments made.
  * A multilayer closure of the incisions will be accomplished using Vicryl sutures.
  Interventions: Device: Patient Specific Titanium Eminoplasty
- Inlay Autogenous Bone Graft (Active Comparator): * A safety distance of 5 mm will be maintained from the apex of the mandibular incisor and inferior mandibular border, the mental foramen, and permanent canine follicle.
  * One corticocancellous bone block with a maximum depth of 4 mm will be removed by mallet and chisel based on the recommendation that bone from the chin should be harvested at this maximum depth, compatible with the course of the mandibular incisive nerve canal on CT scans.
  * After removal of bone from the chin, the intervening bone struts will be removed using rongeur forceps and used as an additional bone graft.
  * The bone removed will be trimmed and contoured in a wedge form to be used as an inter-positional graft in the previously down fractured articular eminence to act as an obstacle in front of the mandibular condyle to prevent its hyper movement.
  Interventions: Procedure: Inlay Autogenous Bone Graft

INTERVENTIONS:
Device: Patient Specific Titanium Eminoplasty — * The stages of virtual surgical planning and fabrication of patient specific titanium eminoplasty will be designed my Mimics 15 program.
  * Once designed, the virtual design and surgery will be planned on a computer model where vital anatomical structures could be identified and thus could be avoided during surgery.
  * After obtaining all the dataset needed from the CT scan, the collected data will be sent to the Egyptian soil, water and environmental institution for manufacturing, packing and sterilization of the patient specific titanium eminence.
  * The patient specific titanium eminence will be inserted and secured with two to three screws of individual lengths according to the virtual plan.
  * Functional mandibular movements were reproduced to confirm absence of subluxation and checked for interference and any required adjustments made.
  * A multilayer closure of the incisions will be accomplished using Vicryl
  Arms: Patient Specific Titanium Eminoplasty
Procedure: Inlay Autogenous Bone Graft — * Steps to harvest the bone graft:
  * Down-fracture of the articular eminence to be augmented with Inlay bone graft to increase the vertical height of the articular eminence. A green-stick fracture will be created avoiding a possible complete fracture of the lower segment of the eminence
  * To obtain Inlay bone graft from the chin, anterior mandibular vestibule incision will provide good access to the mandibular symphysis.
  Arms: Inlay Autogenous Bone Graft

SUMMARY:
In the small and highly specialized field of TMJ surgical treatments, restriction of the mandibular condylar movement outside of the articular eminence is one of the treatment choices suggested in TMJ dislocation.

Limitation of translation of the condyle in TMJ dislocation by inlay autogenous bone graft is the classic method to hinder the movement of the condyle beyond the articular eminence.

Patient specific TMJ prosthesis is very promising nowadays that it will not only build on the strengths of the current TMJ systems but will take advantage of digital innovations in custom design and three-dimensional(3D) printing of TMJ prosthesis. Moreover, TMJ Titanium eminoloplasty was reported to be a predictable and flexible instrument for TMJ dislocation treatment.

Thus, the investigators are conducting this study to compare the effect of both methods on the improvement of the maximal incisal opening of patients with chronic mandibular condylar dislocation, aiming to solve the problem of increasing the mouth opening of patients in their daily mouth opening. Also to reduce the community's fear from such a problem, which sometimes prevent patients from seeking treatment at their dentists leading to more serious complications that can be avoided. Furthermore, the investigators are trying to provide an evidence for oral and maxillofacial surgeons in order to provide the best quality service with the least expenses and thus gaining the patients' trust and saving time, money and effort.

ELIGIBILITY:
Inclusion Criteria:

* Medically free patients.
* Long-standing dislocation of the TMJ for more than 3 weeks and the failure of manual reduction.
* Failure of conservative strategies such as orientation to self-limit jaw movement and the use of a chin-cap or bandage.
* Previous failed TMJ surgery.
* Age range is between 18 and 40 years with no sex predilection.
* Patients who can understand Visual Analogue Scales (VAS) and are able to sign informed consent
* Highly motivated patients

Exclusion Criteria:

* Pregnant females.
* Patients having a significant systemic disorder.
* Psychological disorders, drug or alcohol dependency.
* Known allergies or sensitivities to dental materials, including Titanium or general anasethic agents.
* Severe medical conditions that would not allow management in the clinic.
* Inability to return for follow up visits.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2018-12-01 (Estimated); Primary Completion 2019-12-01 (Estimated); Study Completion 2020-02-01 (Estimated)

PRIMARY OUTCOMES:
The maximal incisal opening | 9 months
  will be measured using a caliper.

IPD SHARING:
Plan to Share IPD: Undecided